CLINICAL TRIAL: NCT05689385
Title: The Effectiveness of eHealth-based Cardiac Rehabilitation in Post-myocardial Infarction Patients：a Randomized Controlled Trial.
Brief Title: eHealth-based Cardiac Rehabilitation in Post-myocardial Infarction Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202207060RINC
Record Dates: First submitted 2023-01-03; First posted 2023-01-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction
Keywords: cardiac rehabilitation; telerehabilitation; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eHealth-based cardiac rehabilitation (Experimental): Participants receive a 12-wk case manager-led eHealth-based cardiac rehabilitation program with follow-up at 12 week, 6 months and 12 months.
  Interventions: Other: eHealth-based cardiac rehabilitation
- Usual care (No Intervention): Participants receive usual care.

INTERVENTIONS:
Other: eHealth-based cardiac rehabilitation — The 12-wk case manager-led eHCR program includes:
  1. Individualized exercise prescription according to the results of cardiopulmonary exercise test.
  2. At least one session of in-person physical therapy to familiarize participants with the process of exercise training before the initiation of telerehabilitation.
  3. Telerehabilitation: a 30-minute moderate aerobic exercise training with remote monitoring and instruction using video conferencing. (Frequency: twice per week in the first 4 weeks, once per week in the 5th-8th week, once every 2 weeks in the 9th-12th week)
  4. Additional self-exercise to achieve the target volume of 150-minute moderate aerobic exercise and 2 sessions of resistance training per week.
  5. Patient education for secondary prevention delivered regularly via a communication app on the smartphone.
  6. Weekly follow-up call from a case manager via phone call or communication app.
  Other Names: eHCR
  Arms: eHealth-based cardiac rehabilitation

SUMMARY:
The goal of this randomized controlled trial is to compare the effect of eHealth-based cardiac rehabilitation with the effect of usual care on exercise capacity and qualify of life in patients after myocardial infarction.

DETAILED DESCRIPTION:
Cardiac rehabilitation can improve exercise capacity, life of quality, readmission rate and mortality rate for patients after myocardial infarction. International guidelines list cardiac rehabilitation after myocardial infarction as class IA recommendation. However, low participation rate of cardiac rehabilitation due to barriers such as lacking of time, transport or affordability issues is an unsolved problem worldwide.

eHealth, consisting of telemedicine, mobile health and personalized care using wearable devices has the potential to remove the barriers and become an effective model to deliver cardiac rehabilitation. Thus, we design a randomized controlled trial to compare the effect of a case manager-led eHealth-based cardiac rehabilitation program with usual care on the compliance, physical activity, quality of life, and cardiorespiratory fitness in patients after myocardial infarction.

ELIGIBILITY:
Inclusion criteria:

1. ≥ 20 years of age.
2. Within 6 months after the onset of acute myocardial infarction.
3. At lowest to moderate risk according to the guideline from American Association of Cardiovascular and Pulmonary Rehabilitation.
4. Unable or refused to attend center-based cardiac rehabilitation.

Exclusion criteria:

1. Unable to walk independently or use a stationary bike.
2. Unable to follow verbal command.
3. Not having a smartphone which can get on the internet.
4. Having contraindications for exercise according to American College of Sports Medicine's Guidelines for Exercise Testing and Prescription.
5. Unable to provide informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change of peak oxygen uptake | at baseline, 12 weeks(post-intervention), and 12 months.
  Peak oxygen uptake will be assessed using cardiopulmonary exercise test before intervention, at 12 weeks (post-intervention), and at 12 months.
Change of ventilatory anaerobic threshold | at baseline, 12 weeks(post-intervention), and 12 months.
  Ventilatory anaerobic threshold will be assessed using cardiopulmonary exercise test before intervention, at 12 weeks (post-intervention), and at 12 months.

SECONDARY OUTCOMES:
Adherence to prescribed exercise | at 12 weeks(post-intervention) and 12 months.
  The degree of completion of prescribed exercise will be assessed at 12 weeks and 12 months.
Evaluation of Quality of life | at baseline, 12 weeks(post-intervention), and 12 months.
  The investigators will assess the change in 36-Item Short Form Survey(SF-36).
Depression | at baseline, 12 weeks(post-intervention), and 12 months.
  The investigators will assess the change in Patient Health Questionnaire (PHQ-9). The PHQ-9 score ranges from 0-27. Higher scores indicate worsen symptoms.
Anxiety | at baseline, 12 weeks(post-intervention), and 12 months.
  The investigators will assess the change in Generalized Anxiety Disorder scale (GAD-7). The GAD-7 score ranges 0-21. Higher scores indicate worsen symptoms.
Evaluation of physical activity | at baseline, 12 weeks(post-intervention), and 12 months.
  The investigators will assess the change in physical activity using Long form International Physical Activity Questionnaire(IPAQ) Taiwan version.
Evaluation of grip strength | at baseline, 12 weeks(post-intervention), and 12 months.
  The grip strength will be measured using a grip goniometer with the participants seated and the elbow flexed at 90 degrees.
Evaluation of isometric knee extension strength | at baseline, 12 weeks(post-intervention), and 12 months.
  The isometric knee extension strength will be measured using a dynamometer with participants seated and knee flexed at 90 degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Jui Chuang, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No